CLINICAL TRIAL: NCT04006691
Title: A Phase 3b Multicenter Extension Trial Evaluating the Efficacy and Safety of UGN-101 (Mitomycin Gel) for Instillation on Ablation of Upper Urinary Tract Urothelial Carcinoma in Recurrent Patients From Trial TC-UT-03
Brief Title: Efficacy and Safety of UGN-101 in Recurrent Patients
Acronym: Retreatment
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to projected low enrollment, it has decided not to move forward with the study.
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-UT-03/E
Record Dates: First submitted 2019-06-12; First posted 2019-07-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma; Transitional Cell Carcinoma; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: TC-3; MitoGel; UGN-101; UTUC; Ureteral; Upper Tract; Carcinoma; Kidney; Renal; Ureter; Gel; Local; Mitomycin C; Prolonged Release; Slow Release; Kidney Sparing; T1; T0; Low Grade; Transitional Cell Carcinoma of Renal Pelvis; TCC
MeSH Terms: conditions — Carcinoma; Carcinoma, Transitional Cell | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-101 instillations (Experimental): The Mitomycin C (MMC) concentration of UGN-101 to be used in this trial will be 4 mg MMC per 1 mL of TC-3 gel, the maximum dose is 15ml. 3-6 once weekly intravesical instillations for the ablation treatment.
  Interventions: Drug: UGN-101 instillations

INTERVENTIONS:
Drug: UGN-101 instillations — Treatment with UGN-101 once weekly for a total of 3-6 times; in a retrograde fashion.
  Other Names: UGN-101; MitoGel™

SUMMARY:
This trial is designed to evaluate the efficacy and safety of UGN-101 administered to the upper urinary tract (UUT) in patients who were treated in Trial TC-UT-03, found to be a complete response (CR) at the Primary Disease Evaluation (PDE) 1 Visit and are subsequently found to have a documented recurrence of low grade (LG) upper tract urothelial carcinoma (UTUC) at follow up (FU).

DETAILED DESCRIPTION:
This is an open-label, single-arm, Phase 3b multicenter extension trial, designed to evaluate the efficacy and safety of UGN-101 administered to the UUT in patients who were treated in Trial TC-UT-03, found to be a CR at the PDE 1 Visit, and are subsequently found to have a documented recurrence of LG UTUC at FU.

Upon signing of informed consent, the patients will undergo their routine ureteroscopy to assess durability. A biopsy will be performed at Visit 0, if appropriate, to confirm evidence of tumor. If a high grade (HG) UTUC is confirmed by biopsy and/or cytology, the patient will be excluded from the retreatment trial. Eligible patients with confirmed LG non-invasive UTUC will be treated with 3 to 6 once-weekly instillations of UGN-101 in a retrograde fashion, per investigator's discretion.

Five weeks (± 1 week) following the last Investigational product (IP) treatment, the patient will be assessed for efficacy and safety at the PDE 2 Visit. At this visit, the patient will undergo ureteroscopy and any remaining lesions will be biopsied, and UUT urine wash will be collected for cytology.

Patients demonstrating CR at the PDE 2 Visit will undergo FU visits at 3, 6, 9, and 12 months (± 2 weeks) following the PDE 2 Visit.

The trial will be approximately 15 months, per patient: a 3- to 6-week treatment period, followed by 4 to 6 weeks post-treatment leading up to the PDE 2 Visit, and a 12-month FU post PDE 2 Visit. This trial will follow the Steering Committee, and a Data Monitoring Committee (DMC) has been assigned as established for the primary trial TC-UT-03.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients with recurrent LG UTUC who were found to be CR at the PDE 1 Visit (in Trial TC-UT-03).
2. Biopsy taken from 1 or more tumors located in the UUT shows LG urothelial carcinoma (up to 2 months before Visit 0). If there are tumors in both the kidney and the ureter, at least 1 biopsy should be taken from each location.
3. Urine wash cytology sampled from the UUT documenting the absence of HG urothelial cancer.
4. Patients must have adequate organ and bone marrow function as determined by routine laboratory tests.
5. Patient has no active urinary tract infection (UTI) as confirmed by urine culture or urinalysis

Main Exclusion Criteria:

1. Patient intends to be treated with systemic chemotherapy during the duration of the trial.
2. Patient with urinary obstruction.
3. Inability to deliver the IP to the UUT.
4. Patient has any other medical or mental condition(s) that make(s) their participation in the trial unadvisable in the opinion of the treating investigator.
5. Patient has a contraindication to mitomycin treatment, or known sensitivity to mitomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | An average of 11 weeks
  Complete response defined dichotomously as "Success" if CR was confirmed at the end of the treatment period (PDE 2 Visit), and "Failure" otherwise.

SECONDARY OUTCOMES:
Long-term durability of complete response (CR) | 3, 6, 9 and 12 months
  This endpoint is defined only for those patients demonstrating CR at the PDE 2 Visit.

OTHER OUTCOMES:
Incidence (number of patients) of adverse events | 15 months
  Adverse events (AEs) analyses will include only Treatment Emergent Adverse Events (TEAEs), namely, those events which started on the day of first trial IP administration or afterwards.
  The incidence (no. of patients) of TEAEs will be provided when broken down by System Organ Class (SOC) and by Preferred Term (PT) according to MedDRA dictionary;
  * Breakdowns of TEAEs by all AEs attributes will also be provided;
  * Breakdowns of TEAEs by age, sex and volume of instillation will also be provided;
  * The incidence of serious TEAEs will be provided when broken down by System Organ Class (SOC) and by Preferred Term (PT) according to MedDRA dictionary as well as by serious adverse events (SAEs) attributes and by age, sex, and volume of instillation. SAEs will also be listed.
Frequency (number of events) of adverse events | 15 months
  Adverse events (AEs) analyses will include only Treatment Emergent Adverse Events (TEAEs), namely, those events which started on the day of first trial IP administration or afterwards.
  The Frequency (no. of patients) of TEAEs will be provided when broken down by System Organ Class (SOC) and by Preferred Term (PT) according to MedDRA dictionary;
  * Breakdowns of TEAEs by all AEs attributes will also be provided;
  * Breakdowns of TEAEs by age, sex and volume of instillation will also be provided;
  * The Frequency of serious TEAEs will be provided when broken down by System Organ Class (SOC) and by Preferred Term (PT) according to MedDRA dictionary as well as by serious adverse events (SAEs) attributes and by age, sex, and volume of instillation. SAEs will also be listed.
Clinically meaningful changes in laboratory values of blood hematology, coagulation, liver and kidney function parameters and urinalysis | 15 months
  Changes from baseline in laboratory values and incidence of measurements defined as Potentially Clinically Significant (PCS) will include the following:
  Complete blood count (CBC, including red blood, cell indices, and white blood cell differential, Platelet count), Creatinine, Blood urea nitrogen, Uric acid, Sodium, Potassium, Phosphorus, Calcium, serum glutamate oxaloacetate transaminase/aspartate aminotransferase (SGOT/AST), serum glutamate pyruvate transaminase/Alanine transaminase (SGPT/ALT), gamma-glutamyl transferase (GGT), Alkaline phosphatase, Total Bilirubin, Direct Bilirubin, Albumin, Total protein, Prothrombin Time and International Normalized Ratio, and Urinalysis (Specific gravity, power of hydrogen (pH), Glucose, Urobilinogen, Bilirubin, Blood, Protein, Nitrites, Leukocyte Esterase, Microscopic examination, Bacteriuria (if required) and White blood cells)
Clinically meaningful changes in vital signs assessments values (blood pressure, pulse and temperature) | 15 months
  Changes from baseline in vital signs assessments values and incidence of measurements of Potential Clinical Significance (PCS) will include blood pressure, pulse, and temperature
Clinically meaningful changes in full physical examination values including General appearance, Cardiovascular and Respiratory system, HEENT (head, eyes, ears, nose, and throat) and neck, Abdomen Extremities, Neurologic system, Skin and Urological system | 15 months
  Any clinically-relevant changes occurring during the trial visit will be recorded in the AE sections of the case report form (CRF). Full general physical examination will be done on visits 0, 7, and 11 Urology-oriented physical examinations will be done on visits 0, 7, 8, 9, 10, and 11.
  Full physical examination findings are composite outcome measure consisting of multiple measures:
  General appearance, Cardiovascular system, Respiratory system, HEENT (head, eyes, ears, nose, and throat) and neck, Abdomen Extremities and Neurologic system Skin
  Urology-Oriented physical examination findings are composite outcome measure consisting of multiple measures:
  Urethral meatus, Perineal skin and mucus membranes Scrotum and testes (for male patients), Lymphadenopathy, Rectal examination (Screening visit only) Bimanual examination (female patients - Screening visit only)

CONTACTS AND LOCATIONS:
Overall Officials: Ifat Klein, Phd, Study Director — UroGen Pharma
Locations (5):
- United States (4):
  - UCLA - University of California, Los Angeles, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - John Hopkins University, Baltimore, Maryland
  - Urology Center Las Vegas, Las Vegas, Nevada
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No